CLINICAL TRIAL: NCT00915122
Title: A Phase I/II Study of Dose Escalated Intensity Modulated Radiation Therapy (IMRT) for the Treatment of Pelvic Lymph Nodes and Primary Tumour in Patients With Carcinoma of the Prostate
Brief Title: Intensity Modulated Radiation Therapy (IMRT) Pelvic Nodes Prostate
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 05-0396-C
Record Dates: First submitted 2009-06-02; First posted 2009-06-05 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: IMRT treatment for Prostate cancer patients; Radiation treatment for prostate cancer; cancer of the prostate; Patients with high risk adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- IMRT in prostate cancer (Experimental)
  Interventions: Radiation: Dose Escalated IMRT

INTERVENTIONS:
Radiation: Dose Escalated IMRT — Patients will receive external beam RT 55.1Gy in 29 once daily fractions to pelvic lymph nodes/prostate/seminal vesicles followed by 24.7Gy in 13 once daily fractions to the prostate/seminal vesicles using intensity modulated radiation therapy.

SUMMARY:
The purpose of this study is to determine the feasibility and late toxicity of dose escalated radiation therapy to the pelvic lymph nodes and prostate and seminal vesicles in the treatment of high risk prostate cancer. All eligible patients with high risk prostate cancer who are going to have primary radiation therapy to the pelvic lymph nodes and prostate seminal vesicles with or without concurrent hormonal therapy will be approached regarding study entry.

DETAILED DESCRIPTION:
Prostate cancer is now the most commonly diagnosed cancer in Canadian men and is the third most common cause of cancer death.1 Locally advanced prostate cancer (clinical T3/T4) is uncommon in North America because of earlier diagnosis following widespread PSA testing and patient information campaigns. However, in the past decade the term high-risk prostate cancer has been developed to include the previous locally advanced disease and patient with T1/T2 disease with poor prognostic features (either a high Prostate Specific Antigen or high Gleason score). The risk of involvement of pelvic lymph nodes by prostate cancer for certain subgroups of intermediate risk and most high risk prostate cancer may be substantial. The long term results of conventional dose (66-70 Gy) external beam radiation therapy for intermediate and locally advanced prostate cancer have been disappointing. The combination of hormonal therapy and radiation therapy or radiation therapy dose escalation are the two strategies which have been evaluated and are now used to improve these results.

ELIGIBILITY:
Inclusion Criteria:

* A histologic diagnosis of adenocarcinoma of the prostate within six months of entry.
* Clinical Stage T1-T2 with (PSA >20 or Gleason score >7)
* Clinical Stage T3, T4
* Bone scan reported as negative for metastases within 6 months of study entry.
* All patients must have a CT scan of the abdomen and pelvis reported as negative for nodal metastases within 12 wks of study entry.
* The patient must not have received greater than 6 months of hormonal therapy.
* The patient must not have received cytotoxic anticancer therapy prior to study entry.
* Patients must have an ECOG performance status of 2 or less.
* Age 80 years old or less
* Signed informed consent

Exclusion Criteria:

* Patients with history of inflammatory bowel disease or other contraindication to radical radiation therapy
* Patients with prior colorectal surgery
* Patients with prior or active malignancy except non-melanoma skin carcinoma within 5 years of the diagnosis of prostate cancer

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2005-11; Primary Completion 2010-09 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility and late toxicity of dose escalated radiation therapy to the pelvic lymph nodes and prostate and seminal vesicles in the treatment of high risk prostate cancer. | after all patients have completed study intervention

SECONDARY OUTCOMES:
acute toxicity of therapy;prostate motion when pelvic radiotherapy is delivered;treatment time required to deliver IMRT to the pelvic lymph nodes, prostate and seminal vesicles | after all patients have completed study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Tara Rosewell, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Bayley A, Rosewall T, Craig T, Bristow R, Chung P, Gospodarowicz M, Menard C, Milosevic M, Warde P, Catton C. Clinical application of high-dose, image-guided intensity-modulated radiotherapy in high-risk prostate cancer. Int J Radiat Oncol Biol Phys. 2010 Jun 1;77(2):477-83. doi: 10.1016/j.ijrobp.2009.05.006. Epub 2009 Sep 3. PMID 19733014